CLINICAL TRIAL: NCT00354146
Title: A Phase 2 Study Evaluating the Efficacy of the Farnesyl Transferase Inhibitor (FTI) R115777 in Patients With Refractory or Relapsed Acute Myeloid Leukemia (AML)
Brief Title: A Phase 2 Study of Farnesyl Transferase Inhibitor (R115777, Tipifarnib) in Patients With Refractory or Relapsed Acute Myeloid Leukemia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR004036
Record Dates: First submitted 2006-07-18; First posted 2006-07-20 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Leukemia, Nonlymphocytic, Acute
Keywords: Farnesyl transferase inhibitor; relapsed or refractory acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — tipifarnib

INTERVENTIONS:
Drug: tipifarnib (R115777)

SUMMARY:
The purpose of this study is to evaluate the effectiveness (response rate) and safety of tipifarnib in patients with refractory or relapsed AML.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) accounts for approximately 25% of all cases of leukemia diagnosed in the Western hemisphere. First-line chemotherapy regimens induce complete remissions in 55-75% of patients. However, between 50% and 70% of patients who achieve remission will relapse. Current therapy for patients refractory to initial therapy or who relapse within 6 months of remission is unsatisfactory because complete remission rates are low and remission duration is brief. New drugs with novel mechanisms of action may be more beneficial than the currently available ones. Tipifarnib represents a new class of oncology drugs which have a specific cellular target (inhibition of the farnesyl transferase protein), one of the components of the Ras oncogene, as its specific mechanism of acton. It is believed that inhibition of this protein will lead to a decrease of cellular proliferation or cell death. This is an open-label, multicenter, non-comparative phase 2 study investigating the efficacy and safety of farnesyl transferase inhibition with tipifarnib administered orally as a single agent, twice daily, for the first 21 days of every 28 day cycle. Patients are enrolled by disease status into two cohorts; Cohort 1 includes patients with relapsed AML and Cohort 2, patients with refractory AML. All patients will be treated for a sufficient length of time to determine response to study medication (effectiveness) by evaluating the rate of complete remission (CR) or complete remission with incomplete platelet recovery (CRp), duration of complete remission, time to disease progression and progression-free survival, overall survival, and to characterize clinical benefit and quality of life (QOL). The safety profile of tipifarnib will also be determined in patients with refractory of relapsed AML.. The patients will receive six tablets (100 mg each) of tipifarnib twice daily for 21 of 28 day cycles (7 day rest period between cycles). Patients may receive tipifarnib until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Refractory or relapsed Acute myeloid leukemia (AML)
* Eastern Cooperative Oncology Group (ECOG) performance of 0-2
* any value of WBC
* able to eat food and medication orally
* females must use contraception and not be pregnant

Exclusion Criteria:

* .Not in another study with an investigational agent within 3 weeks of tipifarnib administration
* must not have active CNS leukemia
* must not have disseminated intravascular coagulation (DIC) disorder with evidence of hemorrhage
* must not be allergic to imidazole drugs such as ketoconazole, miconazole, econazole, or terconazole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2001-04; Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
The objective is to determine the rate of complete remission or complete remission with incomplete platelet recovery induced by tipifarnib in patients with refractory or relapsed AML treated until disease progression or unacceptable toxicity occurs.

SECONDARY OUTCOMES:
These objectives are to determine the objective remission rate, duration of remission, time to disease progression/progression-free survival, overall survival, and the clinical benefit/quality of life (QOL). The safety profile will also be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.